CLINICAL TRIAL: NCT06196528
Title: WristArt Total Wrist Arthroplasty Implant First In Human Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fibioseq Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLN-0001
Record Dates: First submitted 2023-11-26; First posted 2024-01-09 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2023-12

CONDITIONS: Wrist Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- WristArt implantation (Experimental)
  Interventions: Device: WristArt implant

INTERVENTIONS:
Device: WristArt implant — implantation of the WristArt implant

SUMMARY:
The WristArt implant will be implanted for the first time in humans' wrists

ELIGIBILITY:
Inclusion Criteria:

1. Subjects suffering from one the following conditions:

   1. Osteoarthritis (OA) of the wrist joint due to various causes (age, trauma, Avascular Necrosis)
   2. Rheumatoid arthritis of the wrist joint or other rheumatological diseases which destroy the wrist joint
   3. Unrepairable previous intraarticular fractures of the distal radius, scaphoid or lunate bones of the wrist joint (i.e., historical fractures that were failed to fuse surgically)
   4. Symptomatic congenital abnormalities around wrist joint such as carpal bones coalition, mild forms of Madelung's deformities etc.
   5. Patients who underwent failed proximal row carpectomy, or failed partial carpal bones fusion
2. Patients who's their wrist x-ray shows no damage to the carpal bones that are not fused as part of the surgery
3. Patient Rated Wrist Evaluation Score (PRWE) at baseline is above 70 points out of 100
4. Visual Analog Pain Score (VAS) at baseline is above 70 points out of 100

Exclusion Criteria:

1. Patients younger than 18 years old
2. Patients for whom bone growth did not complete yet
3. Paralytic hand patients
4. Patients with sensitivity to Titanium (ADD/CHANGE MATERIALS AS NEEDED)
5. Cerebral palsy patients with wrist joint contracture and loss of sensation in the hand
6. Low quality of capitate bone and/or excessively short capitate bone (≥50% destruction) due to various causes (AVN, comminuted fracture, lytic lesions, congenital etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2024-01-02 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Number of Device Related Serious Adverse events at 6 months post operation | 6 months post operation
  Implantation Safety profile at 6 months post operation
Number of cases with Fully and successfully implanted device at the end of surgery per surgeon's reporting and radiological imaging | 48 hours post-surgery
  Implantation Success profile at the end of surgery

SECONDARY OUTCOMES:
Number of Device Related Serious Adverse events at 24 months post operation | 24 months following implantation
  Implantation Safety profile at 24 months post operation
Average Pain Reduction levels according to Visual Analog Pain Score (VAS) | 1 month, 3 months, 6 months, 1 year, 2 years
  Pain is calculated using a visual analog scale ranges from 1-10 (taken from the pain subscale of the Patient Reported Wrist Evaluation PRWE scale)
Average levels of change in functionality according to Patient Reported Wrist Evaluation (PRWE) | 1 month, 3 months, 6 months, 1 year, 2 years
  The PRWE is a 15-item questionnaire designed to measure wrist pain and disability in activities of daily living. scores range from 0 (no disability) to 100 (worse functional score)
Average levels of change in Grip Strength as measured by dynamometer | 1 month, 3 months, 6 months, 1 year, 2 years
  levels of change in Grip Strength as measured by a dynamometer
Average levels of change in Range of motion as measured by a goniometer | 1 month, 3 months, 6 months, 1 year, 2 years
  levels of change in Range of motion
Implant loosening rate per radiological measurements | 1 month, 3 months, 6 months, 1 year, 2 years
  Implant loosening rate per radiological measurements
Metal Ion Levels in blood at 1 year following surgery | 1 year
  Metal Ion Levels in blood at 1 year following surgery
Average Surgical Satisfaction Questionnaire (SSQ-8) | 1 year
  SSQ8 is a 8-items instrument, with responses recorded on a 5-point Likert-type scale from 0 (worst) to 4 (best) and an overall score ranging from 0 (very unsatisfied) to 32 (very satisfied)
Levels of change in functionality according to quick DASH scores (0 - full function ; 100 - impaired functionality) | 1 month, 3 months, 6 months, 1 year, 2 years
  Levels of change in functionality according to quick DASH scores

CONTACTS AND LOCATIONS:
Overall Officials: Amir Oron, Principal Investigator — Kaplan Medical Center
Locations (1):
- Kaplan Medical Center, Rehovot, Israel

IPD SHARING:
Plan to Share IPD: Undecided